CLINICAL TRIAL: NCT07353242
Title: "THE EFFECT OF BUTEIKO RESPIRATORY TECHNIQUE APPLIED TO ASTHMA PATIENTS ON FATIGUE, EXERCISE CAPACITY, AND ASTHMA CONTROL"
Brief Title: The Effect of Buteyko Breathing Technique on Asthma Patients
Acronym: Buteyko Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Adile Nese, Assos Prof., University of Gaziantep
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Buteyko Breathing Technique
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma,; Buteyko; Fatigue; Breathing Exercises; Exercise Capacity; Asthma Control
MeSH Terms: conditions — Asthma; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Buteyko group (Experimental): In the Buteyko group, in addition to standard treatment, participants received training and practice in the Buteyko Breathing Technique aimed at reducing hyperventilation. The intervention was delivered as face-to-face group training by an internationally certified instructor and included a 30-minute theoretical session followed by practical exercises. These consisted of controlled breath-holding with reduced breathing performed while seated and walking, as well as a relaxation phase focusing on nasal breathing accompanied by calming music. Mouth taping was used throughout the exercises to promote nasal breathing. Participants were instructed to perform the exercises at home three times daily, with weekly outpatient follow-up visits, and were monitored for a total of six weeks.
  Interventions: Other: Buteyko Breathing Technique

INTERVENTIONS:
Other: Buteyko Breathing Technique — This intervention is distinguished by its standardized delivery by an internationally certified Buteyko practitioner and its integration of key Buteyko components, including reduced breathing, controlled breath-holding, nasal breathing with mouth taping, and relaxation. It incorporates both seated and walking-based exercises, uses objective measures such as Control Pause and step counting, and includes a structured home-based practice with weekly follow-up over six weeks.

SUMMARY:
This study was designed as a pre-test-post-test randomized controlled experimental trial to determine the effects of buteyko breathing technique application on fatigue, exercise capacity, and asthma control in asthma patients.The study, planned as a randomized controlled experimental study, included a total of 90 participants.

The sample consisted of asthma patients who applied to the Chest Diseases outpatient clinic of Gaziantep University Application and Research Hospital, had been diagnosed with asthma within the last 6 months, did not have heart failure, did not have communication or perception problems, did not have walking disabilities, and were between 18-59 years old.Following random assignment, participants were divided into two groups of 45 participants each. The groups were: 1) Buteyko 2) Control

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory airway disease that affects individuals of all ages and represents a major public health problem due to its high prevalence and substantial clinical, social, and economic burden. In addition to respiratory symptoms, fatigue and functional limitations are common yet often overlooked in individuals with asthma, significantly impairing daily life. Alongside pharmacological treatments, low-cost, safe, and easily applicable non-pharmacological approaches are gaining increasing importance in asthma management. One such approach is the Buteyko breathing technique, a non-pharmacological breathing retraining method aimed at reducing hyperventilation, improving breathing patterns, and alleviating asthma symptoms. However, evidence regarding the effects of the Buteyko breathing technique on fatigue, functional exercise capacity, and asthma control remains limited. Therefore, this study aims to evaluate the effects of the Buteyko breathing technique on fatigue levels, functional exercise capacity, and asthma control in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with asthma within the last 6 months
* Absence of heart failure
* Absence of communication and perception problems
* Absence of walking impairment Being between 18-59 years of age-

Exclusion Criteria:

* -Child patients
* Those diagnosed with heart failure
* Conditions that impede walking
* Those with communication and perception problems

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
The Asthma Control Test (ACT) | 6 weeks
  The Asthma Control Test (ACT) is a practical, patient-completed scale consisting of five questions, scored between 5 and 25 points, that assesses the level of asthma control; higher scores indicate better control.

SECONDARY OUTCOMES:
The Chronic Obstructive Pulmonary Disease and Asthma Fatigue Scale (COPD) | 6 weeks
  The Chronic Obstructive Pulmonary Disease and Asthma Fatigue Scale (COPD) is a 12-item, five-point Likert-type scale that assesses fatigue in individuals with asthma and COPD; higher scores indicate higher fatigue levels.

CONTACTS AND LOCATIONS:
Overall Officials: Adile Neşe, Study Director — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aluwı, M. F., Azmı, N. A., Zanudın, A., & Ramlı, A. (2025). Effect of Buteyko Breathing Technique and Inspiratory Muscle Training on Acute Exacerbation of Bronchial Asthma in a 55-Year-Old Patient: A Case Report. Buletin SK, 9(1), 55-60
- [Result] AbdElmawla Elsaid, R. A., Zahran, W. E. K., & Elsaid Hafez, D. M. (2023). Comparison of the Effects of Buteyko and Diaphragmatic Breathing Technique on Improving Pulmonary Functions and Asthma Control among Patients with Bronchial Asthma. Egyptian Journal of Nursing and Health Sciences, 4(3), 58-76.
- [Result] Abd Allah Abd El Hafeez, N., Khalil Hafez, M., Mohamed Ahmed, Z., Metwally El-Sayed, M., Abdelwahab Khedr, M., & Fathy Ahmed Dawood, R. (2025). Evaluating the Effect of Buteyko Breathing Technique in Enhancing Asthma Control and Life Quality Among Asthma Patients: A Nursing-Led Quasi-Experimental Study. Egyptian Journal of Health Care, 16(1), 831-852.